CLINICAL TRIAL: NCT04386837
Title: The Inter-rater Reliability of the Turkish Version of Aphasia Rapid Test for Stroke
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Mariam Kavakci, Speech-Language Pathologist Manager, Ankara City Hospital Bilkent
Other Study IDs: AnkaraCHBilkentFTR1
Record Dates: First submitted 2020-05-09; First posted 2020-05-13 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Aphasia
Keywords: stroke; aphasia; reliability
MeSH Terms: conditions — Aphasia; Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aphasics: Patients with a left MCA infarct due to CVA will be included in the study. Each subject will be administered an aphasia screening test less than 3 minutes in length. The same test will be administered by another clinician to the same patient within a maximum of 12 hours to assess the inter-rater reliability of the test.
  Interventions: Other: Turkish Aphasia Rapid Test

INTERVENTIONS:
Other: Turkish Aphasia Rapid Test — Same

SUMMARY:
The Aphasia Rapid Test (ART) is a bedside aphasia screening test developed originally in French. The purpose of this study is to assess the inter-rater reliability of the Turkish version of the ART in stroke patients.

DETAILED DESCRIPTION:
The Aphasia Rapid Test (ART) was developed and validated originally in French to evaluate language skills in post-stroke patients (Azuar et al., 2013). It is a 26-point scale that takes less than 3 minutes to administer. The simplicity of the ART allows it be used bedside in acute post-stroke patients with little to no training needed. The items needed to administer the ART are also easy to access in healthcare settings (e.g., watch, pen, doctor's coat). Although the ART is not a diagnostic test, it is beneficial for tracking progress and determining prognosis in stroke patients.

The original ART was designed similar to the NIH Stroke Scale (NIHSS), a widely-used test in stroke patients. The NIHSS which assesses many areas of functioning (level of consciousness, gaze, visual ability, facial palsy, motor and sensory ability, limb ataxia, language, dysarthria, and extinction and inattention) was chosen because of its sensitivity to early changes in neurological status and high prognostic accuracy (http://www.nihstrokescale.org). The ART is an expanded version of the language section of the NIHSS. The total possible points on the ART is 26, which indicates the highest level of impairment. The test begins with the patient being asked to follow two one-step commands (up to two points each), a complex command (up to 3 points), repeat three nouns (up to 6 points), repeat a simple sentence (up to 2 points), and name three simple objects (up to 6 points). The next item requires a rating of dysarthria by the examiner (up to 3 points). On the final item, the patient is asked to name as many animals as they can think of in one minute (up to 4 points). With the exception of items 1a, 1b, and 6, there are no time restrictions on the test.

The purpose of the present study is to translate the original ART into Turkish to provide an efficient method for the evaluation of language skills in post-stroke Turkish-speaking patients and to assess its inter-rater reliability.

ELIGIBILITY:
Inclusion Criteria:

* Left MCA infarct due to CVA
* Right hand dominant
* Turkish as first language
* CVA within the last 10 days

Exclusion Criteria:

* Right or bilateral brain lesion
* Previous stroke
* Psychiatric disorder
* Other neurological disorder
* Cognitive impairment
* Endotracheal entubation prohibiting responses to test

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of left MCA stroke patients who experienced a CVA within the last 10 days. These patients will consist of males and females with a minimum age of 18.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Inter-rater reliability | The test will be administered within a time frame of 12 hours by two clinicians
  The inter-rater reliability between two clinicians administering the same test

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Kavakci, PhD, Study Director — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kavakci M, Koyuncu E, Tanriverdi M, Adiguzel E, Yasar E. The inter-rater reliability of the Turkish version of Aphasia Rapid Test for stroke. Top Stroke Rehabil. 2022 May;29(4):272-279. doi: 10.1080/10749357.2021.1923314. Epub 2021 Jun 1. PMID 34060434